CLINICAL TRIAL: NCT05431010
Title: Efficacy on Walking Ability of Electroacupuncture Therapy in Elderly Patients with Sarcopenia：a Randomized Controlled Trial
Brief Title: Efficacy on Walking Ability of Electroacupuncture Therapy in Elderly Patients with Sarcopenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Wenzhe Wu, Attending Physician, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022ZB186
Record Dates: First submitted 2022-06-12; First posted 2022-06-24 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Sarcopenia
Keywords: sarcopenia；electroacupuncture; geriatric
MeSH Terms: conditions — Sarcopenia | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- electroacupuncture and rehabilitation training (Experimental): Participants in this group will received electroacupuncture（EA） combined with Otago exercise program(OEP). Acupuncture will be executed with size 0.30×40mm needle. EA will be performed with electronic acupuncture instruments
  Interventions: Device: electroacupuncture; Behavioral: Rehabilitation Training
- rehabilitation training only (Active Comparator): The rehabilitation group will be only treated with the Otago exercise program(OEP). The Otago Exercise is a program developed by the research group of fall prevention in the elderly led by Campbell of Otago Medical University in the 1990s. It is a home exercise program aimed at strengthening lower extremity muscle, balance and preventing falls in the elderly. Otago Exercise combines resistance exercise, balance training and aerobic walking and is an exercise prescription for elderly patients with sarcopenia (details are as follows).
  Interventions: Behavioral: Rehabilitation Training

INTERVENTIONS:
Device: electroacupuncture — Participants are required to be in the supine position. Routine disinfection first. Participants are then subjected to acupuncture and achieve deqi sensation at all acupuncture points. Four paired of acupuncture points (i.e. Biguan acupoints and Futu points; Yanglingquan acupoints and Zusanli acupoints, identical on both sides) are connected to the EA devices. EA parameter is set as sparse wave and frequency is 2Hz. The intensity of the EA is determined by the patients' tolerance. Needles will be left in place and each session of EA will last 30 minutes. Participants will undergo a total of 36 EA sessions, with the frequency of 3 sessions every week for 12 weeks.
  Arms: electroacupuncture and rehabilitation training
Behavioral: Rehabilitation Training — The rehabilitation training group will be only treated with the Otago exercise program(OEP). Otago Exercise combines resistance exercise, balance training and aerobic walking and is an exercise prescription for elderly patients with sarcopenia.
  1. Exercise: including warm-up exercise (5 minutes) + resistance exercise (20 minutes) + balance training (5 minutes). Training intensity: 30 minutes a day, 3 times a week, once every other day, 12 weeks of training period; resistance exercise gradually increases the load.
  2. Walking program: Take a walk. Activity intensity: 30 minutes each time, 2 times a week, combined with exercise (walking during the interval between exercise sessions), 12 weeks of training period

SUMMARY:
Introduction: The efficacy of existing therapies for the treatment of sarcopenia is still not satisfactory. Therefore, this randomized controlled, assessor-blinded study was designed to investigate the efficacy and safety of electroacupuncture(EA) therapy in elderly patients with sarcopenia.

Methods and analysis: This randomized controlled trial will enroll 120 elderly patients with sarcopenia. Subjects will be randomly assigned in a 1:1 ratio to either EA combined with rehabilitation training group or rehabilitation training group through a central computerized randomization system. Primary outcome measure is lower limb mobility, including 6-minute walk test、timed get up and go test, and short physical performance battery. Secondary outcome measures include lower limb muscle mass and lower limb muscle strength. Outcome assessment will be conducted before the intervention, at 12 weeks after the intervention and at the end of the 12-week follow-up. Adverse reactions will be evaluated during the trial.

Conclusion: This research will provide evidence to clarify whether EA is effective and safe in the treatment of sarcopenia.

DETAILED DESCRIPTION:
Introduction: The efficacy of existing therapies for the treatment of sarcopenia is still not satisfactory. Therefore, this randomized controlled, assessor-blinded study was designed to investigate the efficacy and safety of electroacupuncture(EA) therapy in elderly patients with sarcopenia.

Methods and analysis: This randomized controlled trial will enroll 120 elderly patients with sarcopenia. The experimental group is EA combined with rehabilitation training group, while the control group is rehabilitation training group. Rehabilitation training is the more recognized treatment method for sarcopenia all over the world. Eligible subjects will be randomly assigned to two group in a 1:1 allocation ratio. All participants will undergo 12 weeks of treatments in two groups. This protocol is based on the standards for Reporting Interventions in Clinical Trials of Acupuncture (STRICTA) and the SPIRIT reporting guidelines. Primary outcome measure is lower limb mobility, including 6-minute walk test、timed get up and go test, and short physical performance battery. Secondary outcome measures include lower limb muscle mass and lower limb muscle strength, such as lower extremity skeletal muscle mass、appendicular skeletal muscle mass、calf circumference、knee flexion and extension strength and grip strength. Outcome assessment will be conducted before the intervention, at 12 weeks after the intervention and at the end of the 12-week follow-up. Adverse reactions will be evaluated during the trial.

Conclusion: This research will provide evidence to clarify whether EA is effective and safe in the treatment of sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

1. 60 years ≤ age ≤ 95 years, male or female;
2. Patients are able to walk and communicate independently, and can complete required rehabilitation training;
3. Patients meet the diagnostic criteria proposed by the Asian Working Group for Sarcopenia(AWGS);
4. Patients volunteer to participate in this study and sign the informed consent.

Exclusion Criteria:

1. Patients with serious primary diseases of heart, brain, liver, kidney and hematopoietic system;
2. Patients with severe mental illness, cognitive impairment, and disorientation;
3. Patients have trauma and unsuitable for sports;
4. Patients with electronic devices or metal objects implanted in the body;
5. Patients can't complete the required rehabilitation training;
6. Patients cannot receive EA treatment due to any reasons
7. Patients are participating in other drugs, acupuncture and massage trials.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
6min walk test | 12 weeks
  The 6-min walking test setup is a straight line of 20 meters on a flat floor, and a chair is placed at each end as a sign. The subjects walk back and forth between them. The pace of walking is determined according to their own physical fitness, and they walk as fast as possible. In this way, the maximum walking distance that an individual can reach within 6 minutes will be texted
time to get up and go(TGUG) | 12 weeks
  The TGUG test measures the time it takes for an individual to get up from a chair, complete a short 3 meters round-trip walk, and finally sit back in the chair.
short physical performance battery (SPPB) | 12 weeks
  SPPB is a comprehensive test instrument that includes a walking speed test, a sit-to-stand test, and a balance test. The Walking Speed Test measures the time to pass a distance of 4 meters at daily walking speed. Sit-to-stand test is to calculate the time to complete 5 consecutive sets of getting up-sit down. The balance test includes 3 parts: 10 seconds for standing on the left and right side of both feet; standing on half front and half rear feet and standing on front and rear feet

SECONDARY OUTCOMES:
lower extremity skeletal muscle mass | 12 weeks
  The skeletal muscle mass of the lower limbs can be detected separately by applying the BCA body composition analyzer produced by Tsinghua Tongfang
appendicular skeletal muscle mass(ASMM) | 12 weeks
  The BCA body composition analyzer produced by Tsinghua Tongfang can be used to directly test the skeletal muscle mass of the extremities.
calf circumference | 12 weeks
  Measured by applying a measuring tape horizontally around the circumference of the thickest part of the calf
knee flexion and extension strength | 12 weeks
  The TB-ISO multi-joint isometric strength testing system (made in Italy) was applied to test the peak moment/peak moment body weight ratio, average power, and total work for the isometric exercise of knee flexion and knee extension, respectively.
grip strength | 12 weeks
  grip strength was obtained by grip strength measurement

CONTACTS AND LOCATIONS:
Overall Officials: Wenzhe Wu, Master, Study Director — The Third Affiliated hospital of Zhejiang Chinese Medical University; Ming Guo, Doctor, Principal Investigator — Xiyuan Hospital of China Academy of Chinese Medical Sciences; Hantong Hu, Doctor, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University; Hong Gao, Master, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University; Jinkuo Pang, Bachelor, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University; Yanfei Cao, Master, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University; Yiting Zhang, Master, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
no plan

REFERENCES:
- [Derived] Wu W, Huang X, Fang L, Hu H, Han D. Electroacupuncture Plus Exercise for Sarcopenia in Older Adults: Protocol for a Randomized, Controlled, Assessor-Blinded Trial. Clin Interv Aging. 2025 Oct 23;20:1775-1786. doi: 10.2147/CIA.S545035. eCollection 2025. PMID 41164821